CLINICAL TRIAL: NCT06955429
Title: Observational, Prospective, International and Multicenter Clinical Investigation Measuring the Longterm Clinical Performance and Safety of Biodentine™ XP in Patients Treated for Coronal Restorative or Endodontic Dental Indications.
Brief Title: Clinical Investigation Measuring the Long Term Clinical Performance and Safety of Biodentine™ XP in Patients Treated for Coronal Restorative or Endodontic Dental Indications.
Acronym: BIOD XP
Status: Not yet recruiting | Type: Observational
Sponsor: Septodont (Industry)
Collaborators: Axonal-Biostatem (Industry)
Responsible Party: Sponsor
Other Study IDs: BIOD-XP_2024_01; 2024-A01862-45 (Other: ANSM, BIOLOGICAL RESEARCH AND COLLECTIONS (BRC))
Record Dates: First submitted 2025-04-25; First posted 2025-05-02 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-04

CONDITIONS: Dental Restoration, Permanent; Dental Restorations; Endodontic Treatment
Keywords: Dentine restoration; Coronal carious lesions; Restoration of cervical lesion; Restoration of radicular lesion; Pulp capping; Pulpotomy; Apexification; Revitalization; Endodontic treatment; Root; Crown; Pulp; Root perforations; Furcation perforations; Perforating internal resorptions; External resorption; Root-end filling; Permanent dentine restoration; Temporary dentine-enamel restoration; Biodentine; Biodentine XP

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (3):
- Temporary teeth treated in restorative treatment: For temporary teeth treated in restorative treatment arm, the following restoration indications will be found :
  * In the crown
  * Permanent dentine restoration (including under composites or Inlay/Onlay)
  * Enamel restoration for up to 6 months
  * Restoration of deep and/or large coronal carious lesions
  * Restoration of cervical or radicular lesions
  * On the pulp
  * Direct pulp capping
  * Indirect pulp capping
  * Pulpotomy for diagnosed symptoms of reversible pulpitis and irreversible pulpitis where bleeding is controlled within 5 minutes
  Interventions: Device: Dental restorative or endodontic treatment requiring Biodentine XP use
- Permanent (mature or immature) teeth treated in restorative treatment.: For permanent (mature or immature) teeth treated in restorative treatment arm, the following restoration indications will be found :
  * In the crown
  * Permanent dentine restoration (including under composites or Inlay/Onlay)
  * Temporary dentine-enamel restoration (for up to six-months)
  * Restoration of deep and/or large coronal carious lesions
  * Restoration of cervical or radicular lesions
  * On the pulp
  * Direct pulp capping
  * Indirect pulp capping
  * Pulpotomy for diagnosed symptoms of reversible pulpitis and irreversible pulpitis where bleeding is controlled within 5 minutes
  Interventions: Device: Dental restorative or endodontic treatment requiring Biodentine XP use
- Permanent (mature or immature teeth) treated in endodontic treatment.: For permanent (mature or immature) teeth treated in endodontic treatment arm, the following endodontic indications will be found :
  For permanent teeth (immature or mature):
  * Repair of root perforations
  * Repair of furcation perforations
  * Repair of perforating internal resorption
  * Repair of external resorption
  * Root-end filling in endodontic surgery (retrograde filling)
  For immature permanent teeth with necrotic pulp:
  * Apexification
  * Revitalization procedure relying on root canal revascularisation.
  Interventions: Device: Dental restorative or endodontic treatment requiring Biodentine XP use

INTERVENTIONS:
Device: Dental restorative or endodontic treatment requiring Biodentine XP use — In this observational and prospective study, the patients are included since this intervention is schedulded as part of their routine care.

SUMMARY:
The aim of this present study is to collect additional data for the post-marketing follow-up of Biodentine™ XP and measure long-term (up to 10 years) performance and safety of the biomaterial in all its indications.

DETAILED DESCRIPTION:
This clinical investigation is done according to the European Medical Device Regulation (MDR) 2017/745 and is considered as an observational, post-market clinical follow-up study with no additional invasive and cumbersome procedures. Biodentine™ XP has been marketed in the US since 2022 and was launched in Europe in May 2023.

The aim of the study is to collect additional data for the post-marketing follow-up of Biodentine™ XP and measure long-term (up to 10 years) performance and safety of the biomaterial in its coronal restorative and endodontic dental indications.

The investigators participating in the clinical investigation will be general dental surgeron practitioners, with a great experience in restorative and endodontic indications or in pediatric dentistry, also users of Biodentine™.

This Clinical Investigation is an Observational, Prospective, and Multicenter study. This clinical investigation will take place in several investigational centres in France and Belgium.

This Clinical InvestigatioI is a prospective study: Patients will be treated with the study device (according to its CE-marked Instruction For Use), then followed up.

ELIGIBILITY:
Inclusion Criteria:

1. Temporary tooth, from a child ≥ 2 years old, requiring dental restorative treatment with Biodentine™ XP, and/or, Permanent (mature or immature) tooth, from a child or an adult, requiring a dental restorative and/or an endodontic treatment with Biodentine™ XP.
2. Adult patient with a signed informed consent form; For the minor, if in age to understand, an assent is required, and at least one parent or legal representative must consent.
3. Only in France: Subject affiliated or benefiting from a social/health insurance system.

Exclusion Criteria:

1. Patient with one or more documented contraindication to use Biodentine™ XP (Refer to IFU).
2. Inadequate expected tooth lifetime as estimated by the investigator:

   * For a Temporary tooth: high probability of tooth loss within 2 years after treatment with Biodentine™ XP.
   * For a permanent tooth: high probability of tooth loss within 10 years after treatment with Biodentine™ XP.
3. Patient with any systemic disease that may hinder the normal healing process and/or the follow-up.
4. Adult patient under legal protection measures or unable to express his/her consent, and individual deprived of liberty by judicial or administrative decision, as well as individual receiving psychiatric care.
5. Periodontitis (stage 3, 4 or stage 2 grade C).
6. Inability to comply with study procedures.
7. Participation in another interventional clinical investigation that can induce bias in the study results.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Eligible patients are any male and female, adult patients who have undergone one of the following dental treatments using Biodentine™XP respecting the medical device indications.
Sampling Method: Non-Probability Sample
Enrollment: 275 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2036-07-15 (Estimated); Study Completion 2036-07-15 (Estimated)

PRIMARY OUTCOMES:
Success rate of the treatment with Biodentine™ XP based on clinical and radiographic criteria observed | At 2 years post-treatment for temporary teeth (for radiography if required); • At 10 years post-treatment for permanent (mature or immature) teeth.
  Crown and pulp (restoration) Clinical: No pain, no pulpal symptomatology, no abscesses, no swelling, fistula. Positive response to the pulp vitality electric test.
  Radiographic : No radiolucency at the site of treatment & no wideining of desmodontal space (permanent tooth), Root canal development (permanent immature teeth).
  Indications in the root (endodontic) except revitalization Clinical success: No pain, no inflammation, no abscesses, no swelling and/or fistula. Natural motion or mobility ≤ 1mm, Negative periodontal probing (≤ 4 mm) or positive periodontal probing (> 4 mm) Radiographic success: Absence or reduction of radiolucency at the site of treatment.
  Indications in the root (endodontic) only for revitalization:
  Clinical success: No pain, no abscesses, no swelling and/or fistula, Mobility inferior or equal to the initial situation.
  Radiographic success: Absence or reduction of radiolucency at the site of treatment. Root canal development (for permanent immature teeth)

SECONDARY OUTCOMES:
Success rate of the treatment with Biodentine™ XP based on clinical and radiographic criteria observed | 6 months,1 year for temporary teeth; 6 months, 1 year, 2 years and 5 years for permanent (mature or immature) teeth.
  Treatment success based on clinical and radiographic criteria identical to primary endpoint.
Dentin bridge formation presence (only in restorative indications) | At 6 months, 1 year, 2 years post treatment with Biodentine™ XP for temporary teeth (based on X-ray done if required). At 6 months, 1 year, 2 years, 5 years and 10 years post-treatment for permanent (mature or immature teeth)
  Presence of a dentine bridge observed on the radiographic exam (only for restorative indication).
Safety parameters of Biodentine™ XP during the whole duration of the study including the incidence of treatment-emergent adverse events and device deficiencies. | From treatment onset to 10 years for permanent teeth and 2 years for temporary teeth.
  Safety during the study, based on information collected at each visit:
  Adverse events, only those at least possible related to Biodentine™ XP as judged by both sponsor and investigator: nature, number, severity, relationship with Biodentine™ XP and follow up.
  Biodentine™ XP deficiency: nature, number, severity.

OTHER OUTCOMES:
Usability parameters of Biodentine™ XP on the whole procedure, assessed by the dental surgeon practitioner immediately after use, will be evaluated using a questionnaire designed for dentists. | At the initiation of the study, at its 6-month, 1-year, 2-year, 3-year, 4-year anniversary and after inclusion of all patients in the study.
  Usability of Biodentine™ XP (all patient subgroups): completion of usability questionnaire by dental surgeons after using Biodentine™ XP and user summary questionnaire (overall satisfaction, …).

CONTACTS AND LOCATIONS:
Overall Officials: Dr Katia Jedeon, Principal Investigator — Hôpital Rotschild; Pr Marjorie Zanini, Principal Investigator — Hôpital Pitié Salpêtrière; Pr Marie-Agnès Gasqui De Saint Joachim, Principal Investigator — Hôpital HCL lyon; Dr. Alexis Gaudin, Principal Investigator — Cabinet dentaire; Dr Justine Le Clerc, Principal Investigator — CHRU Rennes; Dr Sandrine DAHAN, Principal Investigator — Cabinet dentaire
Locations (6):
- France (6):
  - HCL Lyon, Lyon
  - Cabinet dentaire, Nantes
  - Cabinet dentaire, Paris
  - Hôpital Rotschild, Paris
  - Hôpital Pitié Salpêtrière, Paris
  - CHU Rennes, Rennes

IPD SHARING:
Plan to Share IPD: Undecided